CLINICAL TRIAL: NCT03249090
Title: "PRO-TECT" Patient Reported Outcomes to Enhance Cancer Treatment
Brief Title: Electronic Patient Reporting of Symptoms During Cancer Treatment
Acronym: PRO-TECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of North Carolina (Other); Mayo Clinic (Other); American Society of Clinical Oncology (Other); American Cancer Society, Inc. (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AFT-39
Record Dates: First submitted 2017-08-01; First posted 2017-08-15 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Self-Reporting of Symptoms (Experimental): Patients report symptoms weekly via web or automated telephone system. Email alerts to nurses for severe/worsening symptoms; printouts for clinicians at visits. Evidence based symptom management pathways provided to patients and clinicians.
  Interventions: Other: Patient Self-Reporting of Symptoms
- Usual Care Delivery (Active Comparator): Evidence-based symptom management pathways provided to patients and clinicians
  Interventions: Other: Usual Care Delivery

INTERVENTIONS:
Other: Patient Self-Reporting of Symptoms — At baseline, CRAs will train patients to self-report symptoms and physical functioning weekly for up to a year, with a choice to do so online or via an automated telephone system. Whenever a concerning symptom is reported, an automated "email alert" notification will be sent to the site CRA. The CRA will forward the alert to the responsible clinical nurse (or other covering clinician) and CC the site's Nurse Champion. Within 72 hours, the CRA will document what action(s), if any, were taken by the nurse in response to the alert (entered by the CRA into a form in the PRO-Core system). A symptom report will be printed/generated by the site CRA whenever the patient has a clinic visit and will be given to the oncologist and nurse caring for the patient.
  Arms: Patient Self-Reporting of Symptoms
Other: Usual Care Delivery — Patients receive routine cancer care delivery with no additional systematic monitoring of symptoms
  Arms: Usual Care Delivery

SUMMARY:
The current study is designed to test nationally whether patients' outcomes and utilization of services can be improved through symptom monitoring via patient-reported outcomes between visits.

DETAILED DESCRIPTION:
This is a cluster RCT at approximately 50 sites where randomization will occur in a 1:1 ratio at the site level (not at the individual patient level). Therefore, approximately 25 sites will be randomized to the PRO-TECT intervention arm (patient-reporting of symptoms), and approximately 25 sites will be randomized to the control arm (usual care delivery). Approximately 1200 patients will be enrolled. Specifically:

PROCEDURES AT ALL SITES (CONTROL SITES AND INTERVENTION SITES):

* Site staff (CRA and Nurse Champion required) will attend the site initiation webinar with UNC staff, including training for the PRO-Core online data management system and orientation to the symptom management guidelines.
* At enrollment, all participants will be given a booklet with patient-level symptom advice and a link to the content online.
* All participants will receive compensation for participation, mailed to them as gift cards by UNC.
* CRAs will train all participants how to complete outcomes questionnaires for the trial using the PRO-Core online system. Participants will be given a choice to complete these in clinic or from home online, or if necessary via paper in clinic (with the CRA entering the data into PRO-Core). If the patient does not self-complete this information, the CRA will contact them to collect the information and then enter it into PRO-Core. The outcomes questionnaires will be completed at baseline; and at month 1 (+/- 2 weeks); and at months 3, 6, 9, and 12/off-study (+/- 4 weeks each), and will be available in English, Spanish, or Mandarin Chinese. At each time point, the CRA will contact the participant to remind them about the upcoming questionnaire and offer help.
* Chart abstraction will be conducted by CRAs at baseline and at off-study for each participant, with data entered into the PRO-Core system. Date of death information will additionally be abstracted at 18 and 24 months, and possibly later per the UNC study team.
* CRAs will be asked to complete a feedback survey (entered by the CRA into the PRO-Core online system) and may be asked to participate in a brief telephone debriefing and/or site visit.
* Accrual will be monitored in a weekly teleconference between the UNC team and site CRAs.

ADDITIONAL PROCEDURES AT INTERVENTION SITES ONLY:

* At baseline, CRAs will also train patients to self-report symptoms and physical functioning using the PRO-Core system weekly for up to a year, with a choice to do this online or via an automated telephone system (patient choice), and a choice of English, Spanish, or Mandarin Chinese.
* Whenever a concerning symptom is reported, an automated "email alert" notification will be sent to the site CRA. The CRA will forward the email alert to the responsible clinical nurse (or other covering clinician) and CC the site's Nurse Champion. Within 72 hours, the CRA will document what action(s), if any, were taken by the nurse in response to the alert (entered by the CRA into a form in the PRO-Core system).
* A symptom report will be printed/generated by the site CRA whenever the patient has a clinic visit, and will be given to the oncologist and nurse caring for the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (21+) with metastatic cancer of any type (EXCEPT leukemia or indolent [slow growing] lymphoma)
2. Receiving outpatient systemic cancer treatment for non-curative/palliative intent, including chemotherapy, targeted therapy, or immunotherapy.
3. Enrolled at any point in their treatment trajectory, meaning during any line of treatment, and at any point during a course or cycle of treatment.
4. Can understand English, Spanish, and/or Mandarin Chinese.

Exclusion Criteria:

1. Cognitive deficits that would preclude understanding of consent form and/or questionnaires.
2. Current participation in a therapeutic clinical trial (because these often involve PRO questionnaires and intensive monitoring).
3. Patients being treated with curative intent (e.g., adjuvant chemotherapy for breast, lung, or ovarian cancer; primary curative therapy for testis cancer or lymphoma).
4. Receiving hormonal therapy only (e.g., tamoxifen or aromatase inhibitors in breast cancer; androgen deprivation therapy in prostate cancer; or octreotide in neuroendocrine cancers)
5. Indolent lymphomas (due to their prolonged time courses that may be minimally symptomatic).
6. Leukemias (time courses inconsistent with other tumor types in chronic and acute leukemias).
7. Does not understand English, Spanish, or Mandarin Chinese.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1197 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Basch, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (45):
- United States (45):
  - Grand Valley Oncology, Grand Junction, Colorado
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Eastern Maine Medical Center, Bangor, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Meritus Medical Center, Hagerstown, Maryland
  - Lowell General Hospital, Lowell, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St. Joseph Mercy Ann Arbor Hospital, Ypsilanti, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Mercy Clinic Cancer and Hematology - Chub O'Reilly Cancer Center, Springfield, Missouri
  - Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nevada Cancer Specialists, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - Montefiore Medical Center/ Albert Einstein College of Medicine, The Bronx, New York
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health - York Cancer Center, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - MD Anderson Cancer Center, Houston, Texas
  - Centra Lynchburg Hematology Oncology Clinic, Lynchburg, Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Vincent Hospital Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basch E. Toward patient-centered drug development in oncology. N Engl J Med. 2013 Aug 1;369(5):397-400. doi: 10.1056/NEJMp1114649. Epub 2013 Jul 3. No abstract available. PMID 23822654
- [Background] Reilly CM, Bruner DW, Mitchell SA, Minasian LM, Basch E, Dueck AC, Cella D, Reeve BB. A literature synthesis of symptom prevalence and severity in persons receiving active cancer treatment. Support Care Cancer. 2013 Jun;21(6):1525-50. doi: 10.1007/s00520-012-1688-0. Epub 2013 Jan 12. PMID 23314601
- [Background] Henry DH, Viswanathan HN, Elkin EP, Traina S, Wade S, Cella D. Symptoms and treatment burden associated with cancer treatment: results from a cross-sectional national survey in the U.S. Support Care Cancer. 2008 Jul;16(7):791-801. doi: 10.1007/s00520-007-0380-2. Epub 2008 Jan 17. PMID 18204940
- [Background] Cleeland CS, Zhao F, Chang VT, Sloan JA, O'Mara AM, Gilman PB, Weiss M, Mendoza TR, Lee JW, Fisch MJ. The symptom burden of cancer: Evidence for a core set of cancer-related and treatment-related symptoms from the Eastern Cooperative Oncology Group Symptom Outcomes and Practice Patterns study. Cancer. 2013 Dec 15;119(24):4333-40. doi: 10.1002/cncr.28376. Epub 2013 Sep 24. PMID 24114037
- [Background] Fromme EK, Eilers KM, Mori M, Hsieh YC, Beer TM. How accurate is clinician reporting of chemotherapy adverse effects? A comparison with patient-reported symptoms from the Quality-of-Life Questionnaire C30. J Clin Oncol. 2004 Sep 1;22(17):3485-90. doi: 10.1200/JCO.2004.03.025. PMID 15337796
- [Background] Laugsand EA, Sprangers MA, Bjordal K, Skorpen F, Kaasa S, Klepstad P. Health care providers underestimate symptom intensities of cancer patients: a multicenter European study. Health Qual Life Outcomes. 2010 Sep 21;8:104. doi: 10.1186/1477-7525-8-104. PMID 20858248
- [Background] Atkinson TM, Li Y, Coffey CW, Sit L, Shaw M, Lavene D, Bennett AV, Fruscione M, Rogak L, Hay J, Gonen M, Schrag D, Basch E. Reliability of adverse symptom event reporting by clinicians. Qual Life Res. 2012 Sep;21(7):1159-64. doi: 10.1007/s11136-011-0031-4. Epub 2011 Oct 8. PMID 21984468
- [Background] Fung CH, Hays RD. Prospects and challenges in using patient-reported outcomes in clinical practice. Qual Life Res. 2008 Dec;17(10):1297-302. doi: 10.1007/s11136-008-9379-5. Epub 2008 Aug 18. PMID 18709564
- [Background] Conway PH, Mostashari F, Clancy C. The future of quality measurement for improvement and accountability. JAMA. 2013 Jun 5;309(21):2215-6. doi: 10.1001/jama.2013.4929. No abstract available. PMID 23736730
- [Derived] Stover AM, Deal AM, Ginos B, Dueck A, Spears PA, Jansen J, Carr P, Henson S, Bennett AV, Jonsson M, Snyder C, Basch E. Impact of Providing an Automated Telephone Option to Report Weekly Patient-Reported Outcome Measures in the PRO-TECT Trial (AFT-39) on Disparity Gaps in Symptom Management and Outcomes. JCO Clin Cancer Inform. 2025 May;9:e2500046. doi: 10.1200/CCI-25-00046. Epub 2025 May 23. PMID 40408610
- [Derived] Mody GN, Bennett AV, Stover AM, Jonsson M, Teal R, Vu M, Carda-Auten J, Jansen J, Carr P, Dueck A, Henson S, Basch E. Implementation of Symptom Monitoring With Electronic Patient-Reported Outcomes: Perspectives and Recommendations From Community Oncology Practices (Alliance AFT-39). JCO Oncol Pract. 2025 Dec;21(12):1830-1837. doi: 10.1200/OP-24-00627. Epub 2025 Apr 11. PMID 40215451
- [Derived] Basch E, Schrag D, Jansen J, Henson S, Ginos B, Stover AM, Carr P, Spears PA, Jonsson M, Deal AM, Bennett AV, Thanarajasingam G, Rogak L, Reeve BB, Snyder C, Bruner D, Cella D, Kottschade LA, Perlmutter J, Geoghegan C, Given B, Mazza GL, Miller R, Strasser JF, Zylla DM, Weiss A, Blinder VS, Wolf AP, Dueck AC. Symptom monitoring with electronic patient-reported outcomes during cancer treatment: final results of the PRO-TECT cluster-randomized trial. Nat Med. 2025 Apr;31(4):1225-1232. doi: 10.1038/s41591-025-03507-y. Epub 2025 Feb 7. PMID 39920394
- [Derived] Lee MK, Mitchell SA, Basch E, Mazza GL, Langlais BT, Thanarajasingam G, Ginos BF, Rogak L, Meek EA, Jansen J, Deal AM, Carr P, Blinder VS, Jonsson M, Mody GN, Mendoza TR, Bennett AV, Schrag D, Dueck AC. Identification of meaningful individual-level change thresholds for worsening on the patient-reported outcomes version of the common terminology criteria for adverse events (PRO-CTCAE(R)). Qual Life Res. 2025 Feb;34(2):495-507. doi: 10.1007/s11136-024-03819-5. Epub 2024 Nov 6. PMID 39503942
- [Derived] Basch E, Schrag D, Henson S, Jansen J, Ginos B, Stover AM, Carr P, Spears PA, Jonsson M, Deal AM, Bennett AV, Thanarajasingam G, Rogak LJ, Reeve BB, Snyder C, Bruner D, Cella D, Kottschade LA, Perlmutter J, Geoghegan C, Samuel-Ryals CA, Given B, Mazza GL, Miller R, Strasser JF, Zylla DM, Weiss A, Blinder VS, Dueck AC. Effect of Electronic Symptom Monitoring on Patient-Reported Outcomes Among Patients With Metastatic Cancer: A Randomized Clinical Trial. JAMA. 2022 Jun 28;327(24):2413-2422. doi: 10.1001/jama.2022.9265. PMID 35661856
- [Derived] Basch E, Stover AM, Schrag D, Chung A, Jansen J, Henson S, Carr P, Ginos B, Deal A, Spears PA, Jonsson M, Bennett AV, Mody G, Thanarajasingam G, Rogak LJ, Reeve BB, Snyder C, Kottschade LA, Charlot M, Weiss A, Bruner D, Dueck AC. Clinical Utility and User Perceptions of a Digital System for Electronic Patient-Reported Symptom Monitoring During Routine Cancer Care: Findings From the PRO-TECT Trial. JCO Clin Cancer Inform. 2020 Oct;4:947-957. doi: 10.1200/CCI.20.00081. PMID 33112661

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 52 community oncology practices across 25 states between October 2017 and March 2020. The first participant was enrolled on October 30, 2017 and the last participant was enrolled on March 16, 2020. Enrollment was halted short of the enrollment goal of 1200 participants due the uncertainties of the COVID 19 pandemic.
Pre-assignment Details: 1444 participants were assessed for eligibility and 247 were excluded for the following reasons:
  93 did not meet the inclusion criteria 154 declined to participate (1 not enough time to consent, 36 study would take up too much time, 11 patient too sick, 2 patient functional limitations, 41 did not want to fill out survey, 8 did not want contact between visits, 55 no reason given)
Units Other Than Participants: Practices
Groups:
- ePRO Intervention: Patients report symptoms weekly via web or automated telephone system (electronic patient reported outcomes (ePROs)). Email alerts to nurses for severe/worsening symptoms; printouts for clinicians at visits. Evidence based symptom management pathways provided to patients and clinicians.
- Usual Care Control: Evidence-based symptom management pathways provided to patients and clinicians
  Usual Care Control: Patients receive routine cancer care delivery with no additional systematic monitoring of symptoms
Period: Enrollment
Arm/Group | ePRO Intervention | Usual Care Control
Started | 597; 26 Practices | 600; 26 Practices
Completed | 593; 26 Practices | 598; 26 Practices
Not Completed | 4; 0 Practices | 2; 0 Practices
Not completed — Excluded after randomization for ineligibility | 4 | 2
Period: 3 Month Time Point
Arm/Group | ePRO Intervention | Usual Care Control
Started | 593; 26 Practices | 598; 26 Practices
Completed | 542; 26 Practices | 556; 26 Practices
Not Completed | 51; 0 Practices | 42; 0 Practices
Not completed — Death, hospice, discontinued therapy | 41 | 37
Not completed — Voluntary withdrawal | 6 | 3
Not completed — Changed oncology practice | 4 | 2
Period: 12 Month Time Point
Arm/Group | ePRO Intervention | Usual Care Control
Started | 542; 26 Practices | 556; 26 Practices
Completed | 315; 26 Practices | 368; 26 Practices
Not Completed | 227; 0 Practices | 188; 0 Practices
Not completed — Death, hospice, discontinued therapy | 172 | 175
Not completed — Voluntary withdrawal | 35 | 4
Not completed — Changed oncology practice | 20 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ePRO Intervention | Usual Care Control | Total
Number analyzed (Participants) | 593 | 598 | 1191
Age, Customized [Median (Full Range); unit: years] | 64 [29 to 89] | 62 [28 to 93] | 63 [28 to 93]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 359 | 335 | 694
  Male | 234 | 262 | 496
  Missing | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 39 | 53
  Not Hispanic or Latino | 577 | 557 | 1134
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 13 | 24
  Asian | 2 | 16 | 18
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 99 | 94 | 193
  White | 473 | 452 | 925
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 22 | 27
Education [Count of Participants; unit: Participants]
  1st-8th Grade | 10 | 14 | 24
  9th-11th Grade | 35 | 49 | 84
  High School Graduate/GED | 173 | 187 | 360
  Some College, Associate's Degree, Other Certification | 218 | 203 | 421
  College Degree | 91 | 93 | 184
  Advanced Degree | 65 | 50 | 115
  Missing | 1 | 2 | 3
Urban or Rural Site [Count of Participants; unit: Participants]
  Participants at Rural Site | 154 | 163 | 317
  Participants at Urban Site | 439 | 435 | 874
Difficulty Paying Bills [Count of Participants; unit: Participants]
  Not at all | 260 | 224 | 484
  Not very | 106 | 127 | 233
  Somewhat | 161 | 184 | 345
  Very/extremely | 65 | 61 | 126
  Missing | 1 | 2 | 3
Cancer Type [Count of Participants; unit: Participants]
  Colorectal, anal | 100 | 132 | 232
  Thoracic (Lung, Thyroid, Thymus) | 118 | 110 | 228
  Breast | 97 | 80 | 177
  Gyn (Ovarian, Cervix, Uterine, Vaginal) | 64 | 53 | 117
  Pancreas, Hepatobiliary | 48 | 49 | 97
  Gastroesophageal, Small bowel | 25 | 38 | 63
  Genitourinary Non-prostate (Bladder, Kidney, Testicular, Penile) | 36 | 26 | 62
  Myeloma, Lymphoma | 31 | 31 | 62
  Prostate | 33 | 18 | 51
  Melanoma, Skin | 11 | 21 | 32
  Other (Brain, Sarcoma, Other Soft Tissue, Head/Neck, Unknown Primary) | 30 | 40 | 70
Line of Cancer Therapy [Count of Participants; unit: Participants]
  1st Line | 207 | 237 | 444
  2nd Line | 176 | 192 | 368
  3rd Line | 102 | 89 | 191
  4th Line | 108 | 80 | 188

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Unadjusted Kaplan-Meier estimated survival, based on administrative datasets and practice self-report/medical records.
Time Frame: 24 months
Population: Enrolled eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ePRO Intervention | Usual Care Control
Number analyzed (Participants) | 593 | 598
percentage of participants | 42.0 [38.2 to 46.2] | 43.5 [39.7 to 47.6]

2. Secondary Outcome: Physical Functioning
Description: Physical functioning was measured at the 3 month time point using the European Organisation for Research and Treatment of Cancer QLQ-C30 questionnaire. The QLQ-C30 is a widely used 30 item questionnaire with excellent measurement properties. Physical functioning was assessed via 5 items from the QLQ-C30 which generated a single score on a 0-100 point scale (higher scores are better).
  Mean changes from baseline were measured using the QLQ-C30 at 3 months and compared between arms with a linear combination of parameters from a general linear mixed model. Patients who completed the QLQ C30 at baseline and each follow up time point were categorized as improved on each outcome if their score increased by >/=5 points from baseline; worse if their score decreased by >/=5 points and otherwise as stable.
Time Frame: Month 3
Population: Patients who completed the QLQ C30 measure at the 3 month time point.
Measure: Count of Participants; unit: Participants
Arm/Group | ePRO Intervention | Usual Care Control
Number analyzed (Participants) | 522 | 544
Participants
  Improved Physical Functioning (score increased >/=5 points from baseline) | 227 | 195
  Non-responder for Physical Functioning (score changed <5 points from baseline) | 133 | 147
  Worsened Physical Functioning (score decreased >/=5 points from baseline) | 162 | 202

3. Secondary Outcome: Symptom Control
Description: Symptom control was measured at the 3 month time point using the European Organisation for Research and Treatment of Cancer QLQ-C30 questionnaire. The QLQ-C30 is a widely used 30 item questionnaire with excellent measurement properties. Symptom control was assessed as a composite of 8 QLQ-C30 symptom scale scores on a 0-100 point scale (higher scores are better).
  Mean changes from baseline were measured using the QLQ-C30 at 3 months and compared between arms with a linear combination of parameters from a general linear mixed model. Patients who completed the QLQ C30 at baseline and each follow up time point were categorized as improved on each outcome if their score increased by >/=5 points from baseline; worse if their score decreased by >/=5 points and otherwise as stable.
Time Frame: Month 3
Population: Patients who completed the QLQ-C30 measure at the 3-month time point.
Measure: Count of Participants; unit: Participants
Arm/Group | ePRO Intervention | Usual Care Control
Number analyzed (Participants) | 517 | 543
Participants
  Improved Symptom Control (score increased >/=5 points from baseline) | 195 | 158
  Non-responder for Symptom Control (score changed <5 points from baseline) | 199 | 215
  Worsened Symptom Control (score decreased >/=5 points from baseline) | 123 | 170

4. Secondary Outcome: Health-related Quality of Life
Description: Health-related quality of life was measured at the 3 month time point using the European Organisation for Research and Treatment of Cancer QLQ-C30 questionnaire. The QLQ-C30 is a widely used 30 item questionnaire with excellent measurement properties. Health-related quality of life was assessed as a composite of function and symptom scale scores on a 0-100 point scale (higher scores are better).
  Mean changes from baseline were measured using the QLQ-C30 at 3 months and compared between arms with a linear combination of parameters from a general linear mixed model. Patients who completed the QLQ C30 at baseline and each follow up time point were categorized as improved on each outcome if their score increased by >/=5 points from baseline; worse if their score decreased by >/=5 points and otherwise as stable.
Time Frame: Month 3
Population: Patients who completed the QLQ-C30 measure at the 3-month time point.
Measure: Count of Participants; unit: Participants
Arm/Group | ePRO Intervention | Usual Care Control
Number analyzed (Participants) | 517 | 543
Participants
  Improved Health-related Quality of Life (score increased >/=5 points from baseline) | 191 | 154
  Non-responder for Health-related Quality of Life (score changed <5 points from baseline) | 199 | 229
  Worsened Health-related Quality of Life (score decreased >/=5 points from baseline) | 127 | 160

5. Secondary Outcome: Patient Satisfaction/Communication
Description: Patients in the ePRO arm were measured via Patient Satisfaction Questionnaire assessing comprehension of ePRO questions, usability of digital ePRO system, meaningfulness/relevance of ePRO questions, communication/actionability with care team, clinical utility of ePRO system and patient self efficacy. The number of patients analyzed is the number of patients who completed the questions. Some questions were not administered to all patients.
Time Frame: Month 3
Population: Patients participating in the ePROs arm completed the Patient Feedback Survey to assess patient satisfaction with the system and communication with their care team.
Measure: Number; unit: participants
Arm/Group | ePRO Intervention | Usual Care Control
Number analyzed (Participants) | 505 | 0
participants
  Patients who strongly or somewhat agree that ePRO survey questions were easy to understand | 480 |
  Patients who strongly or somewhat agree that the ePRO system was easy to use | 472 |
  Patients who strongly or somewhat agree the ePRO survey questions were relevant to them: number analyzed (Participants) | 392 | 0
  Patients who strongly or somewhat agree the ePRO survey questions were relevant to them | 359 |
  Patients who strongly or somewhat agree the process improved discussions with their care team: number analyzed (Participants) | 504 | 0
  Patients who strongly or somewhat agree the process improved discussions with their care team | 365 |
  Patients who strongly or somewhat agree that their doctor/nurse used the symptom information: number analyzed (Participants) | 502 | 0
  Patients who strongly or somewhat agree that their doctor/nurse used the symptom information | 353 |
  Self-reporting symptoms weekly from home made them feel more in control of their care: number analyzed (Participants) | 504 | 0
  Self-reporting symptoms weekly from home made them feel more in control of their care | 387 |
  Patients who strongly or somewhat agree they would recommend the ePRO system to other patients | 452 |

6. Secondary Outcome: Emergency Department Utilization
Description: Data for emergency department visits were obtained from data abstracted at each practice from the electronic medical record.
Time Frame: 1 year
Population: Enrolled eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | ePRO Intervention | Usual Care Control
Number analyzed (Participants) | 593 | 598
Participants
  No (0) ED Visits | 315 | 273
  1+ ED Visits | 278 | 325

ADVERSE EVENTS:
Time Frame: Participants were assessed for death for up to 2 years.
Description: Dates of death were based on US National Death Index administrative data and confirmed with medical chart abstraction. Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- ePRO Intervention: Patients report symptoms weekly. Email alerts to nurses for severe/worsening symptoms; printouts for clinicians at visits. Evidence-based symptom management pathways provided to patients and clinicians.
- Usual Care Control: Evidence-based symptom management pathways provided to patients and clinicians. Usual Care Control: patients receive routine cancer care delivery with no additional systematic monitoring of symptoms.
Arm/Group | ePRO Intervention | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 350/593 | 345/598
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was conducted during the pandemic when research and clinical resources at participating sites were strained with frequent turnover of staff. This disrupted accrual and conduct and likely decreased the effect size observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT03249090/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT03249090/SAP_001.pdf